CLINICAL TRIAL: NCT03905031
Title: Defining The Operating Characteristics of Near-Infrared Spectroscopy (NIRS) in The Diagnosis of Pediatric Traumatic Intracranial Hemorrhage
Brief Title: Defining the Operating Characteristics of NIRS in the Diagnosis of Pediatric Traumatic Intracranial Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dayton Children's Hospital (Other)
Responsible Party: Principal Investigator, Shobhan Vachhrajani, MD, PhD, FRCSC, Director of Surgical Research, Dayton Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-002
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Craniocerebral Injuries; Head Injuries; Head Injury, Minor; Head Trauma; Traumatic Brain Injury; Traumatic Brain Hemorrhage; Hematoma of Head; Intracranial Hemorrhages
Keywords: Trauma; Traumatic Brain Injury; Infrascanner; Near-Infrared Spectroscopy; Pediatric
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Brain Hemorrhage, Traumatic; Intracranial Hemorrhages; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- InfraScanner 2000 (Experimental): All participants entered into the study will undergo at least one cranial scanning using the InfraScanner 2000 within 4 hours before or after CT scan. Patients will know the results of the CT scan but not of the InfraScanner 2000. A CT result that is positive for hematoma will be considered a true positive and a CT result that is negative for hematoma will be considered a true negative.
  Interventions: Device: InfraScanner 2000

INTERVENTIONS:
Device: InfraScanner 2000 — The InfraScanner is a portable screening device that measures lateralized differences in optical density (OD) to determine the presence of intracranial hematoma. A difference in OD>0.2 is abnormal and suggestive of intracranial hematoma.

SUMMARY:
In this study, investigators look at a different type of technology that might help to avoid having to perform CT scans in certain patients suspected of having a head injury. Near-infrared spectroscopy (NIRS) uses a specific light wavelength to determine if there is bleeding into the head as a result of trauma. Investigators will study NIRS, using a device called the Infrascanner model 2000, to determine if it is as good at detecting bleeding in the head as CT scan, which is the current gold standard. Investigators will try to determine if NIRS can rule in or rule out bleeding into the head, and perhaps this can help to avoid subjecting these youth to the potentially harmful effects of radiation. Investigators will also study how easy it is to use NIRS so that it might become a standard part of the workup for children with suspected head injury.

DETAILED DESCRIPTION:
Patients that present to Dayton Children's Hospital with a head CT order for suspected TBI will be approached for enrollment. An alert will notify study personnel as CT scans are ordered. The goal is to obtain NIRS data within four-hours before or after the CT scan. Informed consent will be obtained according to institutional protocols. NIRS data will be obtained using Infrascanner model 2000 (Infrascanner Inc.). Eight data points will be collected for each subject in standard fashion from right to left frontal, temporal, parietal, and occipital locations. Study personnel will be trained by the manufacturer and will be blinded to the results of the CT scan. Data stored on the Infrascanner will be subsequently transferred to a password-protected database for storage and analysis. For each participant scanned with the Infrascanner 2000, they will be de-identified with a subject number, with patient demographics, mechanism of injury, GCS presentation, time of CT scan, and time of NIRS recorded. CT scan results comprise presence of epidural hematoma and/or subdural hematoma and its maximal thickness if present; presence of intraparenchymal hematoma; presence of skull fracture; and any other traumatic injuries contained in the CT scan report. The length of time required to acquire NIRS data will also be recorded for quality improvement purposes.

The specific aims of this study are to better understand the epidemiology of traumatic brain injury (TBI) at Dayton Children's Hospital, to establish the operating characteristics of NIRS for suspected traumatic intracranial hemorrhage at Dayton Children's Hospital, and to study the implementation of a new diagnostic modality in a busy tertiary care emergency department.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years old
* Glasgow Coma Score (GCS) 3-15
* Undergoing head CT scan for suspected TBI

Exclusion Criteria:

* Post-operative patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of NIRS Optical Density Measurement | Within 4 hours before or after CT scan
  Determine the sensitivity of the NIRS optical density measurement by the Infrascanner device for identifying the presence of intracranial hematomas in pediatric patients after suspected traumatic brain injury compared to head CT scans as the gold standard.
Specificity of NIRS Optical Density Measurement | Within 4 hours before or after CT scan
  Determine the specificity of the NIRS optical density measurement by the Infrascanner device for identifying the presence of intracranial hematomas in pediatric patients after suspected traumatic brain injury compared to head CT scans as the gold standard.
Predictive Values of NIRS Measurement | Within 4 hours before or after CT scan
  Determine the positive and negative predictive values of the NIRS measurements for detecting intracranial hematomas.

SECONDARY OUTCOMES:
Implementation of NIRS in Emergency Department Workflow | 1 year
  NIRS integration into patient care workflow will be measured by surveying those involved in NIRS data acquisition monthly, as well as conducting interviews and focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shobhan Vachhrajani, MD, PhD, Principal Investigator — Dayton Children's Hospital
Locations (1):
- Dayton Children's Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No